CLINICAL TRIAL: NCT04971746
Title: An Open-label, Fixed-sequence Drug-drug Interaction Study in Healthy Subjects to Evaluate the Effect of GLPG4716 on the Pharmacokinetics of Nintedanib and Pirfenidone
Brief Title: Drug-drug Interaction Study with GLPG4716 and Nintedanib and Pirfenidone in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GLPG4716-CL-101; 2021-001718-12 (EudraCT Number)
Record Dates: First submitted 2021-07-20; First posted 2021-07-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-06

CONDITIONS: Healthy
MeSH Terms: interventions — pirfenidone; nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GLPG4716 and pirfenidone (Experimental)
  Interventions: Drug: Pirfenidone; Drug: GLPG4716
- GLPG4716 and nintedanib (Experimental)
  Interventions: Drug: GLPG4716; Drug: Nintedanib

INTERVENTIONS:
Drug: Pirfenidone — On Days 1 and 13, participants will receive an oral dose of pirfenidone.
  Arms: GLPG4716 and pirfenidone
Drug: GLPG4716 — From Day 3 to Day 14, participants will receive GLPG4716 daily.
Drug: Nintedanib — On Days 1 and 13, participants will receive an oral dose of nintedanib.
  Arms: GLPG4716 and nintedanib

SUMMARY:
The main aim of this study is to investigate the possible effect of GLPG4716 on the pharmacokinetics (PK) of pirfenidone and nintedanib. Further aims are to investigate safety and tolerability of GLPG4716 alone or administered simultaneously with pirfenidone or nintedanib.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years of age (extremes included), on the date of signing the informed consent form (ICF). Female subjects should be of non-childbearing potential.
* A body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive.
* Judged to be in good health by the investigator based upon the results of a medical history, physical examination, vital signs, electrocardiogram (ECG), and fasting clinical laboratory safety tests. Aspartate transaminase and alanine aminotransferase must be no greater than the upper limit of normal (ULN). Other clinical laboratory safety test results must be within the reference ranges or test results that are outside the reference ranges need to be considered not clinically significant in the opinion of the investigator

This list only includes the key inclusion criteria.

Exclusion Criteria:

* Known hypersensitivity to ingredients of GLPG4716, pirfenidone, or nintedanib or history of a significant allergic reaction to ingredients of GLPG4716, pirfenidone, or nintedanib as determined by the investigator.
* Treatment with any medication (including over-the-counter (OTC) and/or prescription medication, dietary supplements, nutraceuticals, vitamins and/or herbal supplements, and hormonal replacement therapy) except occasional paracetamol (maximum dose of 2 g/day and maximum of 10 g/2 weeks) in the last 2 weeks or 5 half-lives of the drug, whichever is longer, prior to the first dosing.

This list only includes the key exclusion criteria.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of pirfenidone | From Day 1 pre-dose until Day 15
  To determine the effect of GLPG4716 on the PK of pirfenidone
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) of pirfenidone | From Day 1 pre-dose until Day 15
  To determine the effect of GLPG4716 on the PK of pirfenidone
Cmax of nintedanib | From Day 1 pre-dose until Day 15
  To determine the effect of GLPG4716 on the PK of nintedanib.
AUC0-inf of nintedanib | From Day 1 pre-dose until Day 15
  To determine the effect of GLPG4716 on the PK of nintedanib.

SECONDARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events (SAEs), and TEAEs leading to treatment discontinuations. | From Day 1 through study completion, an average of 2 months
  To evaluate the safety and tolerability of GLPG4716 alone or when co-administered with pirfenidone or nintedanib.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Rueda-Rincon, MD, Study Director — Galapagos NV
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No